CLINICAL TRIAL: NCT00101426
Title: Safety and Efficacy of AS-3201 in the Treatment of Diabetic Sensorimotor Polyneuropathy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sumitomo Pharma Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AS-3201-253
Record Dates: First submitted 2005-01-10; First posted 2005-01-11 (Estimated); Last update posted 2008-01-14 (Estimated); Status verified 2008-01

CONDITIONS: Diabetic Neuropathy
Keywords: Diabetic sensorimotor polyneuropathy; Diabetic Neuropathy
MeSH Terms: conditions — Diabetic Neuropathies | interventions — ranirestat

INTERVENTIONS:
Drug: ranirestat, (AS-3201)

SUMMARY:
This is a safety and efficacy trial of ranirestat(AS-3201) which is an aldose reductase inhibitor in patients with diabetic sensorimotor polyneuropathy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with the following may enter:

Clinical signs and symptoms (footpain, numbness, tingling, weakness, etc.) of symmetrical distal Diabetic Sensorimotor Polyneuropathy with diagnosis by Nerve Conduction Tests and/or Quantitative Sensory Test.

* 18 to 70 years old of either sex and any race
* Type I or Type II, insulin-dependent or non insulin-dependent diabetes for at least six months prior to study entry
* Healthy in general
* No hospitalizations for diabetic control or episodes of ketoacidosis for three months prior to screening
* Female patients of childbearing potential must have a negative serum pregnancy test

Exclusion Criteria:

* Known non-diabetic causes of neuropathic symptoms
* Diabetic patients with no neuropathy or severe neuropathy
* Used any Aldose Reductase Inhibitors within one year of screening
* Clinically significant illness including unstable cardiac, pulmonary, hematologic, hepatic, renal, or neoplastic disease
* A history of systemic carcinoma within five years of screening
* A history of epilepsy or serious head injury
* A history or evidence of drug or alcohol abuse
* Test positive at screening for hepatitis B surface antigen or hepatitis C antibody or have a history of a positive result, or patients with evidence of significant hepatic insufficiency
* A history of known or suspected diagnosis of AIDS, or have tested seropositive for HIV antibody or antigen previously

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500
Dates: Start 2004-10; Study Completion 2006-09

PRIMARY OUTCOMES:
Efficacy

SECONDARY OUTCOMES:
Safety

CONTACTS AND LOCATIONS:
Locations (1):
- Toronto General Hospital, University Health Network, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Bril V, Hirose T, Tomioka S, Buchanan R; Ranirestat Study Group. Ranirestat for the management of diabetic sensorimotor polyneuropathy. Diabetes Care. 2009 Jul;32(7):1256-60. doi: 10.2337/dc08-2110. Epub 2009 Apr 14. PMID 19366965